CLINICAL TRIAL: NCT03952117
Title: Transcranial Direct Current Stimulation of the Motor Cortex in Essential Tremor : A Randomized Controlled Pilot Study
Brief Title: Transcranial Direct Current Stimulation of the Motor Cortex in Essential Tremor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Rechdi Ahdab, M.D , PhD, Lebanese American University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LAUMCRH.RA3.11/Apr/2019
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Essential Tremor; Transcranial Direct Current Stimulation
Keywords: primary motor cortex
MeSH Terms: conditions — Essential Tremor | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCs (Active Comparator): Active tDCS will be administered through a pair of conductive rubber electrodes covered by saline soaked sponges (35 cm2). The current will be delivered continuously at 2 mA for 30 min through a battery-driven constant-current stimulator. The cathode will be positioned facing the primary motor cortex area and the anode over the contralateral supraorbital area.
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham stimulation will be delivered to the motor cortex using a sham tDCS device that delivers a direct current for 10 seconds at the beginning and end of tDCS to provide sensory experiences similar to active stimulation.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS will be administered through a pair of conductive rubber electrodes covered by saline soaked sponges (35 cm2). The current will be delivered continuously at 2 mA for 30 min through a battery-driven constant-current stimulator (Sooma Oy, Helsinki, Finland).

SUMMARY:
The current research is aimed at using Transcranial Direct Current Stimulation (tDCS) as complementary therapeutic tool in the treatment of essential tremor. Patients will be randomized into two groups (tDCS-cathode vs. tDCS-sham) according to detailed protocol. Main outcome will be measured by the change in tremor amplitude using an accelerometer pre and post cathodal tDCS of the motor cortex.

A total of 40 patients ought to be enrolled as specified in methodology. Secondary outcomes will assess TRG essential tremor rating assessment scale (TETRAS) as well as clinical monitoring.

DETAILED DESCRIPTION:
Essential tremor (ET) is a common progressive neurological disorder and is the most common movement disorder. Worldwide , up to 5% of the population suffer from this disorder with an increased incidence with advanced age.

The proposed mechanism that underlies ET, the central oscillating network, is mainly composed of the olivocerebellar system, thalamus and motor cortex. An interruption in this circuit limits the ability of the cortex to reorganize and restore ET. a case of 76 year old female with essential tremor that disappeared following a cortico-subcortical prerolandic stroke despite complete motor recovery highlights the role of the motor cortex in the production and possible therapeutic role of the transcranial direct current stimulation.

Study design A randomized, sham-controlled, double blind and crossover study.

Study procedure:

The first visit is an inclusion visit Prior to starting the first tDCS session, the patient will be asked to fill his/her first TRG essential tremor assessment (TETRAS) scale. The physician will then quantitatively analyze the tremor on the most affected side using an accelerometer. Cathodal tDCS will be administered on the area representing the primary motor cortex and the anode over the contralateral supraorbital area. tDCS stimulation (cathodal and sham) will be done daily for 5 consecutive days during weeks 1 and 5. Each stimulation session will last 30 minutes. tDCS will be performed while the patient is at rest, without any concurrent cognitive or motor task.The two tDCS sessions will be separated by a 23 day washout period.

Patient will be asked to fill out their TETRAS at days 1 and 5 of each tDCS session (cathodal and sham), and days 12 and 19 after each tDCS session (cathodal and sham).

Accelerometer assessment of the tremor will be performed at days 1 and 5 of each tDCS stimulation session (cathodal and sham).

ELIGIBILITY:
Inclusion Criteria:

- Patients who fulfil the 2017 Movement society concusses statement criteria for essential tremor

Exclusion Criteria:

* Isolated focal tremor (voice, head)
* Orthostatic tremor with a frequency of more than 12 Hz
* Task and position specific tremor
* Sudden onset and stepwise deterioration of tremor
* History of substance abuse or dependence in the past
* Co-morbid medical conditions capable of producing or enhancing tremors
* Use of a medication with potential effect on tremor
* History of neurological disorders, brain tumors, brain surgery or abnormal neurological examination
* Epileptic disorders
* Cardiac pacemakers
* Metallic hardware in the head or scalp (surgical clips)
* Eczema or skin abrasion at the intended site of stimulation
* Currently pregnant or plan for pregnancy in the next 6 months
* Patients with prior experience with tDCS
* Major psychosocial problems or medical problems rendering informed consent impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Tremor amplitude | 5 days
  Change in tremor amplitude using an accelerometer pre and post cathodal tDCS of the motor cortex.

SECONDARY OUTCOMES:
Functional impact of tremor | 19 days
  Assess change from baseline of the functional impact of tremor using the TETRAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Rechdi Ahdab, Principal Investigator — Lebanese American University Medical Center
Locations (1):
- LAUMCRH, Beirut, Lebanon

DOCUMENTS (1):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03952117/Prot_000.pdf